CLINICAL TRIAL: NCT01322789
Title: Safety and Efficacy of Mesenchymal Stem Cells in Newly-diagnosed Type 1 Diabetic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Júlio Cesar Voltarelli, Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCFMRPUSP 2; CNPQ 552266/2005-1 (Other Grant/Funding Number: CNPQ 552266/2005-1)
Record Dates: First submitted 2010-12-07; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes mellitus; Stem cells; Autologous stem cell transplantation; Autoimmune diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous mesenchymal stem cell (Experimental): This group wil receive 8 intravenous infusions of mesenchymal stem cells. Four infusions 1 week apart and 4 infusions a month apart
  Interventions: Biological: Intravenous Mesenchymal stem cell infusion

INTERVENTIONS:
Biological: Intravenous Mesenchymal stem cell infusion — Four consecutive intravenous infusions 1 week apart followed by 4 consecutive infusions 1 month apart

SUMMARY:
Type 1 diabetes mellitus results from the autoimmune destruction of the insulin producing pancreatic β-cells. The autoimmune response begins months or even years before the presentation of hyperglycemic symptoms. Previous studies with other autoimmune diseases or acute inflammatory diseases testing the effect of the infusion of mesenchymal stem cells showed promising results in regulating immune system and promoting some degree of disease control. The aim of our study is to determine the safety and efficacy of intravenous infusions of mesenchymal stem cells in newly diagnosed type 1 diabetic patients.

DETAILED DESCRIPTION:
Patients from 12 to 35 years old with type I diabetes mellitus proved by anti-pancreatic beta cell antibodies and recently diagnosed (less than 6 weeks) will be included in this study. First, bone marrow derived adult mesenchymal stem cells are collected from a first degree relative and cultured. After that, the patient receive 4 intravenous infusions 1 week apart followed by 4 infusion 4 months apart.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus diagnosed by clinical/metabolic parameters and positive anti-GAD antibodies
* Less than 6 weeks from diagnosis

Exclusion Criteria:

* Previous diabetic ketoacidosis
* Pregnancy
* Severe psychiatric disorder
* Severe organic impairment (renal, hepatic, cardiac, pulmonary)
* Active infectious disease
* Previous or present neoplastic disease

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-09; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
AUC C-peptide levels during mixed meal tolerance test | pré-treatment, 6 months, 12 months and then yearly (course of study 7 years)
Safety | Every 6 months until death
  The process of analyzing safety data is made daily based on clinical interview, frequent physical examination and general laboratory findings weekly from the first stem cell infusion until 60 months after the last infusion. Chest X-ray will be performed in days 100, 180, 270, 360 after the lest infusion and then every 6 months. Fecal occult blood, alpha pheto protein, beta-human chorionic gonadotropin, carcino-embrionary antigen, abdomen ultrasound will be performed in month 6 and 12 after the last infusion and then yearly.

SECONDARY OUTCOMES:
Daily insulin use | Daily (course of study is 7 years)
Hemoglobin A1C | 3 months
Anti-GAD titres | Every 6 months
Immunologic reconstitution parameters | Yearly (course of study is 7 years)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Voltarelli, MD, PhD, Principal Investigator — University Hospital, School of Medicine of Ribeirão Preto, Brazil; Carlos E Couri, MD, PhD, Study Chair — University Hospital, School of Medicine of Ribeirão Preto, Brazil
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil